CLINICAL TRIAL: NCT05137639
Title: Free Skin Grafting to Reconstruct Donor Sites After Radial Forearm Flap Harvesting: A Prospective Study With Platelet-rich Fibrin (PRF)
Brief Title: Free Skin Grafting to Reconstruct Donor Sites After Radial Forearm Flap Harvesting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 143/20-me
Record Dates: First submitted 2021-11-12; First posted 2021-11-30 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2021-11

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRF group (Experimental): Participants received platelet-rich fibrin (PRF) prior to free skin grafting
  Interventions: Procedure: Platelet-rich fibrin (PRF)
- non-PRF group (No Intervention): Standard surgical procedure (free skin grafting to reconstruct donor sites without PRF).

INTERVENTIONS:
Procedure: Platelet-rich fibrin (PRF) — PRF was only applied in the experimental arm to improve wound bed conditions
  Arms: PRF group

SUMMARY:
Reconstruction of the donor site after radial forearm flap harvesting is a common procedure in maxillofacial plastic surgery. Unfortunately, free skin graft transplantation faces wound healing impairments such as necrosis, (partial) graft loss, or tendon exposure. Several studies have investigated methods to reduce these impairments and demonstrated improvements if the wound bed is optimized. However, these methods are device-dependent, expansive, and time-consuming. Therefore, the application of platelet-rich fibrin (PRF) to the wound bed could be a simple, cost effective, and device-independent method to optimize wound-bed conditions instead. In this study, PRF membranes were applied between the wound bed and skin graft.

DETAILED DESCRIPTION:
Reconstruction of the donor site after radial forearm flap harvesting is a common procedure in maxillofacial plastic surgery. It is normally carried out with split-thickness or full-thickness free skin grafts. Unfortunately, free skin graft transplantation faces wound healing impairments such as necrosis, (partial) graft loss, or tendon exposure. Several studies have investigated methods to reduce these impairments and demonstrated improvements if the wound bed is optimized, for example through negative pressure wound therapy or vacuum-assisted closure. However, these methods are device-dependent, expansive, and time-consuming. Therefore, the application of platelet-rich fibrin (PRF) to the wound bed could be a simple, cost effective, and device-independent method to optimize wound-bed conditions instead. In this study, PRF membranes were applied between the wound bed and skin graft. Growth factor release could stimulate fibroblast migration, wound healing and angiogenesis. Further more PRF act as a lubricant layer to protect skin graft from tendon motion. This could improve graft in-growth.

ELIGIBILITY:
Inclusion Criteria:

* >18 years, donor site on the forearm after radial forearm flap surgery, free skin graft reconstruction of this skin defect, informed consent

Exclusion Criteria:

* <18 years, inclusion criteria were not met

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Coverage rate | 10-14 days
  The coverage rate was measured 10-14 days after surgery with a photo analysis

SECONDARY OUTCOMES:
Evaluation Score (ES) | 10-14 days
  ES included surgical complications (infection, graft loss..) and was obtained 10-14 days after surgery. Minimum value: 0, maximum value 6. A higher score indicates a worse surgical outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Anton Straub, MD, Principal Investigator — Dep. of Oral and Maxillofacial Plastic Surgery
Locations (1):
- University Hospital of Würzburg, Würzburg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No